CLINICAL TRIAL: NCT04698772
Title: Patient Satisfaction With Subdissociative Dose Ketamine Versus Morphine for Emergency Department Pain Control
Status: Completed | Type: Observational
Sponsor: CHRISTUS Health (Other)
Responsible Party: Principal Investigator, Rebekka Lee, DO, Principal Investigator, CHRISTUS Health
Other Study IDs: 2019-081
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Abdominal Pain
Keywords: Emergency Department; Moderate to severe pain
MeSH Terms: conditions — Abdominal Pain; Emergencies | interventions — Ketamine; Morphine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survey Packet 1 Group: Patients who receive "Packet 1" will be in group 1, or the treatment group. In this packet will be 4 forms: the consent to participate in the study form, a pre-treatment questionnaire (VAS and other demographic information), post-treatment questionnaire (various questions, including demographic questions [age, sex, race, height, weight, etc.], a 10cm (100mm) VAS for pain, a 10cm (100mm) VAS to measure patient satisfaction, and a Likert Scale to measure patient satisfaction), and a form with specific instructions for the physicians to follow that vary depending on whether the instructions are from "Packet 1" or "Packet 2." The physician will be asked to administer a sub-dissociative dose of ketamine for pain control (0.3 mg/kg IV over 3-5 minutes).
  Interventions: Drug: Ketamine
- Survey Packet 2 Group: Patients who receive "Packet 2" will be in group 2, or the control group. In this packet will be 4 forms: the consent to participate in the study form, a pre-treatment questionnaire (VAS and other demographic information), post-treatment questionnaire (various questions, including demographic questions [age, sex, race, height, weight, etc.], a 10cm (100mm) VAS for pain, a 10cm (100mm) VAS to measure patient satisfaction, and a Likert Scale to measure patient satisfaction), and a form with specific instructions for the physicians to follow that vary depending on whether the instructions are from "Packet 1" or "Packet 2."The physician will be asked to administer morphine 4 mg IV push over 3-5 minutes for pain control.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Ketamine — Blinded study group will receive ketamine for pain control (0.3 mg/kg IV over 3-5 minutes)
  Groups: Survey Packet 1 Group
Drug: Morphine — Blinded study group will receive morphine 4 mg IV push over 3-5 minutes for pain control
  Groups: Survey Packet 2 Group

SUMMARY:
The proposed research will be a single blinded (patient) randomized controlled prospective trial of adult patients receiving treatment for moderate to severe abdominal pain to test the hypothesis that patient satisfaction with pain control with Ketamine will be comparable to patient satisfaction with pain control using morphine when treating abdominal pain.

DETAILED DESCRIPTION:
Informed consent will be obtained from patients presenting with chief complaint of moderate to severe abdominal pain in the emergency department who do not meet any exclusion criteria and who willingly agree to participate by signing the written consent form. Investigators will assess the patient's opioid tolerance by asking if they have use an opioid medication in the last week, prescription opioid use at home, and/or recreational opioid use. Patients in both groups will fill out the pre-treatment questionnaire, which will include demographic questions (age, sex, race, height, weight, etc.), a 10cm (100mm) VAS for pain, a 10cm (100mm) VAS to measure patient satisfaction, and a Likert Scale to measure patient satisfaction. Post-treatment survey will be given at 30 minutes after administration of medication. The physician will record whether the patient required additional pain medication after the 30 minutes, final emergency department diagnosis, and final emergency department disposition.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Initial presenting complaint of moderate to severe abdominal pain (five or higher on numerical rating scale [NRS]).
* Subjects will be enrolled into the project one (1) time only.

Exclusion Criteria:

* Under 18 years of age
* Pregnant patients
* Inability to provide written consent
* Evidence of traumatic brain injury
* Hemodynamic instability
* Procedures involving laryngeal manipulation
* History of laryngeal spasm
* History of adverse reaction to Ketamine or morphine
* Patients will not be excluded if they had received pain medications prior to enrollment (ie. Received pain medication from triage, non-physician provider (NPP), or emergency medical services (EMS) prior to being seen by physician
* History of opioid use in the last week, prescription opioid use, recreational opioid use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study subjects include patients presenting to the Emergency Department at CHRISTUS Spohn Shoreline Hospital during a 24 month time frame. Eligible patients will be treated for acute abdominal pain.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
Compare satisfactory scores | 24 months
  The primary outcome parameter is to compare satisfaction scores between patients treated with morphine vs ketamine respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Rebekka Lee, DO, Principal Investigator — CHRISTUS Health
Locations (1):
- CHRISTUS, Corpus Christi, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigator has interest in pursuing future collaboration and grant opportunities.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Background] Morris B, Jahangir A, Sethi, M. Patient Satisfaction: An Emerging Health Policy Issue. AAOS. June 2013. http://www.aaos.org/news/aaosnow/jun13/advocacy5.asp
- [Background] Francis, J. (2018). U.S. Hospitals That Provide Superior Patient Experience Generate 50 Percent Higher Financial Performance Than Average Providers, Accenture Finds. [online] Businesswire.com. Available at: https://www.businesswire.com/news/home/20160511005122/en/U.S.-HospitalsProvide-Superior-Patient-Experience-Generate [Accessed 13 Nov. 2018].
- [Background] "HospitalHCAHPS." CMS.gov Centers for Medicare & Medicaid Services, 21 Dec. 2017, www.cms.gov/Medicare/Quality-Initiatives-Patient-AssessmentInstruments/HospitalQualityInits/HospitalHCAHPS.html.
- [Background] Berkowitz B. The Patient Experience and Patient Satisfaction: Measurement of a Complex Dynamic. Online J Issues Nurs. 2016 Jan 31;21(1):1. doi: 10.3912/OJIN.Vol21No01Man01. PMID 27852212
- [Background] Baker DW. The Joint Commission's Pain Standards: Origins and Evolution. Oakbrook Terrace, IL: The Joint Commission; 2017
- [Background] Axeen S, Seabury SA, Menchine M. Emergency Department Contribution to the Prescription Opioid Epidemic. Ann Emerg Med. 2018 Jun;71(6):659-667.e3. doi: 10.1016/j.annemergmed.2017.12.007. Epub 2018 Jan 16. PMID 29373155
- [Background] Butler MM, Ancona RM, Beauchamp GA, Yamin CK, Winstanley EL, Hart KW, Ruffner AH, Ryan SW, Ryan RJ, Lindsell CJ, Lyons MS. Emergency Department Prescription Opioids as an Initial Exposure Preceding Addiction. Ann Emerg Med. 2016 Aug;68(2):202-8. doi: 10.1016/j.annemergmed.2015.11.033. Epub 2016 Feb 11. PMID 26875061
- [Background] Nsc.org. (2018). Prescription Drug Abuse. [online] Available at: https://www.nsc.org/home-safety/safety-topics/opioids [Accessed 13 Nov. 2018].
- [Background] Motov S, Drapkin J, Likourezos A, Beals T, Monfort R, Fromm C, Marshall J. Continuous Intravenous Sub-Dissociative Dose Ketamine Infusion for Managing Pain in the Emergency Department. West J Emerg Med. 2018 May;19(3):559-566. doi: 10.5811/westjem.2017.12.36174. Epub 2018 Mar 8. PMID 29760856
- [Background] Karlow N, Schlaepfer CH, Stoll CRT, Doering M, Carpenter CR, Colditz GA, Motov S, Miller J, Schwarz ES. A Systematic Review and Meta-analysis of Ketamine as an Alternative to Opioids for Acute Pain in the Emergency Department. Acad Emerg Med. 2018 Oct;25(10):1086-1097. doi: 10.1111/acem.13502. Epub 2018 Jul 17. PMID 30019434
- [Background] Bowers KJ, McAllister KB, Ray M, Heitz C. Ketamine as an Adjunct to Opioids for Acute Pain in the Emergency Department: A Randomized Controlled Trial. Acad Emerg Med. 2017 Jun;24(6):676-685. doi: 10.1111/acem.13172. Epub 2017 Mar 22. PMID 28177167
- [Background] Pourmand A, Mazer-Amirshahi M, Royall C, Alhawas R, Shesser R. Low dose ketamine use in the emergency department, a new direction in pain management. Am J Emerg Med. 2017 Jun;35(6):918-921. doi: 10.1016/j.ajem.2017.03.005. Epub 2017 Mar 2. PMID 28285863
- [Background] Sin B, Tatunchak T, Paryavi M, Olivo M, Mian U, Ruiz J, Shah B, de Souza S. The Use of Ketamine for Acute Treatment of Pain: A Randomized, Double-Blind, Placebo-Controlled Trial. J Emerg Med. 2017 May;52(5):601-608. doi: 10.1016/j.jemermed.2016.12.039. Epub 2017 Mar 6. PMID 28279542
- [Background] Motov S, Rosenbaum S, Vilke GM, Nakajima Y. Is There a Role for Intravenous Subdissociative-Dose Ketamine Administered as an Adjunct to Opioids or as a Single Agent for Acute Pain Management in the Emergency Department? J Emerg Med. 2016 Dec;51(6):752-757. doi: 10.1016/j.jemermed.2016.07.087. Epub 2016 Sep 29. PMID 27693070
- [Background] Motov S, Rockoff B, Cohen V, Pushkar I, Likourezos A, McKay C, Soleyman-Zomalan E, Homel P, Terentiev V, Fromm C. Intravenous Subdissociative-Dose Ketamine Versus Morphine for Analgesia in the Emergency Department: A Randomized Controlled Trial. Ann Emerg Med. 2015 Sep;66(3):222-229.e1. doi: 10.1016/j.annemergmed.2015.03.004. Epub 2015 Mar 26. PMID 25817884
- [Background] Sin B, Ternas T, Motov SM. The use of subdissociative-dose ketamine for acute pain in the emergency department. Acad Emerg Med. 2015 Mar;22(3):251-7. doi: 10.1111/acem.12604. Epub 2015 Feb 25. PMID 25716117
- [Background] Beaudoin FL, Lin C, Guan W, Merchant RC. Low-dose ketamine improves pain relief in patients receiving intravenous opioids for acute pain in the emergency department: results of a randomized, double-blind, clinical trial. Acad Emerg Med. 2014 Nov;21(11):1193-202. doi: 10.1111/acem.12510. PMID 25377395
- [Background] Galinski M, Dolveck F, Combes X, Limoges V, Smail N, Pommier V, Templier F, Catineau J, Lapostolle F, Adnet F. Management of severe acute pain in emergency settings: ketamine reduces morphine consumption. Am J Emerg Med. 2007 May;25(4):385-90. doi: 10.1016/j.ajem.2006.11.016. PMID 17499654
- [Background] Smith DC, Mader TJ, Smithline HA. Low dose intravenous ketamine as an analgesic: a pilot study using an experimental model of acute pain. Am J Emerg Med. 2001 Oct;19(6):531-2. doi: 10.1053/ajem.2001.27152. No abstract available. PMID 11593484
- [Background] Gurnani A, Sharma PK, Rautela RS, Bhattacharya A. Analgesia for acute musculoskeletal trauma: low-dose subcutaneous infusion of ketamine. Anaesth Intensive Care. 1996 Feb;24(1):32-6. doi: 10.1177/0310057X9602400106. PMID 8669651
- [Background] Linking quality to payment. Medicare.gov. https://www.medicare.gov/hospitalcompare/linking-quality-to-payment.html. Published 2018. Accessed November 21, 2018.
- [Background] Rau J. Medicare To Begin Basing Hospital Payments On Patient-Satisfaction Scores. Kaiser Health News. https://khn.org/news/medicare-hospital-patient-satisfaction/. Published 2018. Accessed November 21, 2018.
- [Background] Patanwala AE, Edwards CJ, Stolz L, Amini R, Desai A, Stolz U. Should morphine dosing be weight based for analgesia in the emergency department? J Opioid Manag. 2012 Jan-Feb;8(1):51-5. doi: 10.5055/jom.2012.0096. PMID 22479885